CLINICAL TRIAL: NCT06177522
Title: A Single-arm, Single-center, Exploratory Study of Adebrelimab Combined With Chemotherapy for Neoadjuvant Therapy in Resectable Pancreatic Cancer
Brief Title: Adebrelimab Combined With Chemotherapy for Neoadjuvant Therapy in Resectable Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sizhen Wang, associate chief physician, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZQH-KYLL-23-2601
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab combined with chemotherapy administration group (Experimental): Adebrelimab is a humanized anti-PD-L1 monoclonal antibody independently developed by Hengrui Pharmaceutical. It can block the PD-1/PD-L1 pathway leading to tumor immune tolerance through specific binding of PD-L1 molecules, and reactivate the anti-tumor activity of the immune system, so as to achieve the purpose of tumor treatment.
  Interventions: Drug: Adebrelimab; Drug: albumin-bound paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Adebrelimab — 1200mg，i.v. , q3w
Drug: albumin-bound paclitaxel — 125 mg/m2, i.v.,d1,d8, q3w
Drug: Gemcitabine — 1.0 g/m2, i.v.,d1, d8, q3w

SUMMARY:
Clinical Study on the Safety and Efficacy of the efficacy and safety of Adebrelimab combined with chemotherapy for neoadjuvant treatment of resectable pancreatic cancer

DETAILED DESCRIPTION:
The goal of this clinical trial is to observe and evaluate the efficacy and safety of Adebrelimab combined with chemotherapy for neoadjuvant treatment of resectable pancreatic cancer.The main questions it aims to answer are:

To investigate the feasibility of immunotherapy combined with chemotherapy in the neoadjuvant therapy of pancreatic cancer.

To explore more effective neoadjuvant therapies for pancreatic cancer. Participants will receive 2 cycles of Adebrelimab in combination with albumin-bound paclitaxel and gemcitabine in the neoadjuvant phase, followed by surgery.

ELIGIBILITY:
inclusion criteria

1. Age 18-80 years old, gender unlimited;
2. Patients with resectable pancreatic adenocarcinoma confirmed by histopathology or cytology (CA19-9 > 150 U/ml);
3. No previous systemic treatment for pancreatic cancer;
4. Measurable lesions defined by RECIST standard v1.1 (according to Recist 1.1 standard, the CT scan diameter of tumor lesions is ≥10 mm, and the scan layer thickness is not more than 5 mm);
5. ECOG score: 0 ~ 1;
6. Having adequate organ and bone marrow function, as defined below: Hemoglobin ≥9.0 g/dL neutrophil absolute count ≥1.5×109/L Platelet count ≥100×109/L INR≤1.5 Total bilirubin (TBL) ≤1.5× upper limit of normal (ULN) AST and ALT≤2.5×ULN Serum albumin ≥3.0 g/dL serum creatinine ≤1.5×ULN or measured creatinine clearance > 60 mL/min or creatinine clearance > 60 mL/min calculated according to the Cockcroft-Gault formula (using actual body weight) : Men: creatinine clearance =(weight x (140- age))/(72 x serum creatinine) Women: Creatinine clearance =(body weight x (140-age))/(72 x serum creatinine)x 0.85, where CL=mL/min; Serum creatinine =mg/dL;
7. Patients with active HBV infection should receive antiviral therapy for more than 2 weeks according to local antiviral treatment guidelines before enrollment, and should continue treatment for 6 months after study drug therapy;
8. A negative hepatitis C virus (HCV) antibody test at screening, or a positive HCV antibody test at screening and a subsequent negative HCV RNA test;
9. Expected survival ≥12 weeks;
10. The investigator determined that the patient could receive adabilimab therapy;
11. Subjects voluntarily participate in this study and sign informed consent.

exclusion criteria

1. Concurrent with other uncured malignant tumors;
2. Subjects who have previously used PD-1/PD-L1 antibodies;
3. Subjects who can be surgically resected or treated with radical radiation;
4. Subjects with a history of bleeding and any bleeding event with a severity rating of 3 or above on CTCAE4.0 within 4 weeks prior to screening;
5. Urine routine indicated urinary protein ≥++ and confirmed 24-hour urinary protein quantity > 1.0g;
6. Subjects with poorly controlled hypertension;
7. Subjects who have experienced serious infection within 4 weeks prior to the first dose, including but not limited to infection complications requiring hospitalization, bacteremia, severe pneumonia, etc. Subjects who developed a severe active infection requiring intravenous antibiotic treatment during screening;
8. Subjects requiring systemic treatment with corticosteroids (>10 mg/ day of prednisone or equivalent) or other immunosuppressants within 14 days prior to initial medication. In the absence of active autoimmune disease, inhaled or topical corticosteroids are permitted, as well as adrenal hormone replacement therapy at doses > 10 mg/ day of prednisone efficacy;
9. History of chronic autoimmune diseases, such as systemic lupus erythematosus, ulcerative enteritis, Crohn's disease and other inflammatory bowel diseases; Except for hypothyroidism that requires only hormone replacement therapy and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis or alopecia);
10. Subjects with grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥450 ms for men and ≥470 ms for women). Subjects with NYHA standard Ⅲ ~ Ⅳ cardiac insufficiency or LVEF (left ventricular ejection fraction) < 50% were excluded;
11. Subjects who are preparing for or have previously received tissue/organ transplants;
12. Subjects who have received or will receive live vaccine within 30 days prior to the first dose;
13. Subjects with a history of difficult to control mental illness or severe intellectual or cognitive impairment;
14. Subjects with active hepatitis: hepatitis B virus surface antigen (HBV) positive with HBV DNA≥ 2000 IU/mL, hepatitis C virus antibody (HCV Ab) positive, HCV RNA positive, abnormal liver function, combined with hepatitis B and hepatitis C co-infection;
15. Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
16. Allergic to the experimental drug;
17. Women who are pregnant, breastfeeding or have given birth but refuse to use contraceptives;
18. Other conditions deemed unsuitable for inclusion by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 removal rate | one year
  To observe and evaluate the efficacy and safety of adbelizumab combined with chemotherapy for neoadjuvant treatment of resectable pancreatic cancer
pCR rate | one year
  To observe and evaluate the efficacy and safety of adbelizumab combined with chemotherapy for neoadjuvant treatment of resectable pancreatic cancer

CONTACTS AND LOCATIONS:
Overall Officials: Xinbo Wang, MD, Study Director — Jinling Hospital, China
Locations (1):
- Wang Sizhen, Nanjing, Jiangsu, China